CLINICAL TRIAL: NCT00165971
Title: Recovery From General Anesthesia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: CogState Ltd. (Industry)
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Prevention
Other Study IDs: 459-2003; 19907000
Record Dates: First submitted 2005-09-09; First posted 2005-09-14 (Estimated); Last update posted 2007-04-17 (Estimated); Status verified 2007-04

CONDITIONS: Anesthesia, General; Recovery Period, Anesthesia
Keywords: Cognitive decline; Inflammation; Monitoring; Recovery; Bispectral index
MeSH Terms: conditions — Cognitive Dysfunction; Inflammation

INTERVENTIONS:
Procedure: BIS monitoring

SUMMARY:
General anesthesia allows people to have surgery without experiencing the procedure or pain. To remain unconscious, the depth of sleep must be monitored. Various monitors have been developed, one of which is BIS (short for bispectral index). BIS monitors the level of sleep during anesthesia and improves patient recovery because the amount of sleep drugs can be fine-tuned to the individual. Patients who need a lot to stay asleep get more, and those who need less get less. As a result, patients tend to wake up faster with BIS monitoring as compared to standard practice not using BIS. Little is known about the long-term effects of BIS monitoring. This study investigates whether BIS monitoring during anesthesia improves long-term outcome, well after surgery is over. The hypothesis is that it does. Two groups of patients are compared: one in which BIS monitoring was used, and one in which it was not. Groups are compared on tests of memory, concentration and mental well-being, to see if one does and feels better than the other. The investigators also take blood samples to see how well patients' bodies deal with the surgery. The investigators expect the BIS monitoring group to do better.

DETAILED DESCRIPTION:
Monitoring the effect of sedative drugs, used to anesthetize people during surgery, is complex. Technological advances that focus on brain activity (electroencephalogram, EEG) recently yielded promising parameters, such as the bispectral index (BIS). BIS is a scale from 100 (awake) to 0 (complete cortical EEG suppression), and values between 45 and 60 are recommended for surgical anesthesia. Compared to standard practice, the use of BIS speeds emergence and early recovery from anesthesia while reducing anesthetic drug use. Little is known about the long-term effects of BIS monitoring but it is not unlikely that early improvements in clinical outcome persist over time. Studies have associated first-year postoperative mortality to prolonged periods of too deep surgical anesthesia, as defined by BIS levels below 45. BIS monitoring could thus serve an important function in enhancing patient management and care. Prospective, randomized controlled clinical trials of BIS monitoring and its long-term effects are lacking, however.

The primary goal of this study is to assess whether monitoring of sedation level during general anesthesia, using BIS, enhances long-term recovery. Two outcome domains are of interest: Cognitive function (attention, vigilance, and memory) and immune system responses (inflammation). The former is measured using a computerized test battery while blood samples (cytokines and TNF-a levels) address the latter. Patients are randomly assigned to one of two monitoring groups. While BIS is recorded in both, the values are not available to guide drug dosing in the standard practice group (i.e., blinded). In this group, parameters such as changes in respiration, heart beat, and blood pressure guide the amount of drugs being administered. In the other group, BIS readings are available and used to titrate drugs to values between 50 and 60 (target 55). The anesthetic protocol is similar for both. Recovery is assessed repeatedly in all patients at various intervals after surgery (6 hrs, 1st and 2nd day, and 1 month follow-up). In this way, we intend to capture outcome-variation over time.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing elective hip or knee replacement surgery, primary or revisions, under general anesthesia

Exclusion Criteria:

* Drug allergies
* Recent illicit drug abuse
* Mental illness, or psychoactive medication treatment
* Head trauma resulting in loss of consciousness
* Neurological disorder
* Scheduled for cardiac surgery
* Memory disorders
* Severe visual or auditory handicap
* English is not the patient's first language
* Illiteracy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100
Dates: Start 2003-12; Study Completion 2007-02 (Actual)

PRIMARY OUTCOMES:
Cognitive function
Inflammation

SECONDARY OUTCOMES:
Memory function
Depression
Anxiety

CONTACTS AND LOCATIONS:
Overall Officials: Peter S Sebel, MB BS, PhD, Principal Investigator — Emory University; Chantal Kerssens, PhD, Study Director — Emory University
Locations (1):
- Emory University Hospital, Atlanta, Georgia, United States